CLINICAL TRIAL: NCT05115682
Title: Time of Day Specific Glycaemic and Metabolic Response to High-Intensity Interval Training
Brief Title: Circadian Rhythm and Metabolic Effects of Exercise
Acronym: HITMet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Harriet Wallberg, Prof. MD PhD, Karolinska Institutet
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HIT Metabolome
Record Dates: First submitted 2021-10-19; First posted 2021-11-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2; Circadian Rhythm; Glycemic Control
Keywords: Type 2 Diabetes; High-intensity Intermittent Exercise; Circadian Rhythm; Glycemic Control; Energy Metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: The study will include a group of individuals with type 2 diabetes and a group of individuals with normal glucose tolerance. Each group of participants will complete either a morning (09:00) or an afternoon (16:00) exercise bout. After a one-week washout period, the participants will complete an additional exercise bout at the opposing time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morning First (Experimental): Participants will complete a single bout of exercise at 09:00, and after at least a one-week washout perform another exercise bout at 16:00.
  Interventions: Behavioral: High-intensity Intermittent Exercise
- Afternoon First (Experimental): Participants will complete a single bout of exercise at 16:00, and after at least a one-week washout perform another exercise bout at 09:00.
  Interventions: Behavioral: High-intensity Intermittent Exercise

INTERVENTIONS:
Behavioral: High-intensity Intermittent Exercise — The participants will perform a low-volume, High-intensity Intermittent Exercise bout on a cycle ergometer. Peak exercise capacity of the study participants will be determined on a separate occasion using a ramp-up maximal oxygen consumption test (VO2peak). A single exercise bout will consist of a 7-minute warm-up on a cycle ergometer, followed by 6 1-minute intervals of cycling at individual maximal capacity and 75rpm (rotations per minute). These intervals will be interspersed with 1-min breaks of cycling at low resistance and 75rpm, and the session will conclude with a 3-minute cool-down interval (20 minutes in total).

SUMMARY:
Physical exercise is efficacious in controlling blood glucose levels in individuals with Type 2 diabetes. An individual's exercise capacity and ability to utilize glucose as an energy source oscillates throughout the day. Hence, the beneficial effects of exercise on blood glucose levels may depend on the time of day when the exercise bout is performed. However, the time of day in which the most beneficial adaptations to exercise can be achieved remains unknown. This project aims to answer the following questions: Does time of day impact the beneficial effects of exercise on blood glucose? If so, when can the most beneficial effects of exercise be achieved? Which metabolic mechanisms links time of day, exercise and blood glucose control? To address these questions, individuals with or without Type 2 diabetes will perform an exercise session at two different times (09:00 and 16:00), and continuous glucose monitoring will be used to assess the effects of exercise on blood glucose. We will determine the specific metabolic processes which promote the most beneficial blood glucose response. To achieve this, we will measure which metabolic substrates (carbohydrates, lipids and proteins) are used and which metabolites produced in blood, skeletal muscle and adipose tissue in response to exercise at different times of the day.

DETAILED DESCRIPTION:
Exercise has well-established metabolic benefits and is a preferred intervention for Type 2 diabetes prevention and management. Metabolic determinants of exercise such as skeletal muscle and whole-body substrate oxidation capacity, glucose tolerance and insulin sensitivity and adipose tissue fatty acid release all show circadian oscillations. These rhythms may promote substantially different responses depending on the time of day when exercise is performed.

This is an exploratory study aiming to determine whether exercise at specific times of day can amplify the beneficial effects on glycemia and metabolism in two groups of individuals: those without diabetes or those with Type 2 diabetes (n=40 per group). The primary objective is to determine the glycemic response to an exercise bout at two distinct times of day, measured by continuous glucose monitoring, in men and women with or without Type 2 diabetes. The secondary aim is to identify specific metabolites which facilitate the strongest glycemic response to exercise by examining the whole-body and peripheral tissue metabolomic response to an exercise bout.

The primary goal of the study is to examine the glycemic and metabolic response to exercise within-group for participants with or without Type 2 diabetes. Further comparisons will be made between groups with with or without Type 2 diabetes, across sexes, and by individual chronotype (determined by a standardized questionnaire) to examine the variation in the exercise response across these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI): 23 - 33 kg/m2
* Participants diagnosed with Type 2 Diabetes (insulin independent) or participants without Type 2 Diabetes (based on normal HbA1c and fasting glucose levels).
* Ability to provide informed consent
* Ability to complete the exercise regiment

Exclusion Criteria:

* Medications: Insulin
* Current nicotine user (cigarettes, snus, nicotine gum) or past nicotine users less than 6 months before inclusion in the study
* Pre-existing cardiovascular condition (Angina pectoris, Cardiac arrhythmia, Cardiac infarction, Coronary stent / angiography, Cerebrovascular insult, Hypertension [> 160 mmHg systolic, or > 95 mmHg diastolic])
* Pre-existing blood-borne disease (HIV, Hepatitis C, MRSA)
* Pre-existing systemic or localized rheumatic illness
* Malignant Disease
* Pre-existing psychiatric disorder
* Another pre-existing systemic disease

Ages: 45 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Exercise-induced Changes in 24 Hour Interstitial Glucose Concentration | 3 days (1 day before to 1 day after exercise)
  Glucose excursions will be charted using continuous interstitial glucose monitors. The day immediately before exercise will be used as baseline, the day of exercise to assess the acute response, and the day after exercise to assess lasting effects on glycemia. Exercise effects on glucose concentration will be primarily assessed by comparing 24-hour curves between conditions.

SECONDARY OUTCOMES:
Acute Exercise-induced Changes in Interstitial Glucose Concentration | 2 hours (0 minutes before to 120 minutes after exercise)
  Glucose will be charted using continuous glucose monitors. Acute response to exercise, during the exercise bout and during an additional 120 minutes will be compared between conditions.
Interstitial Glucose Concentration Response to a Meal | 2 days (1 day before and day of exercise)
  Glucose will be charted using continuous glucose monitors. Three standardized meals per day will be provided on each occasion for the day before, day of and day after exercise. The 120 minute glucose response to the standardized meal succeeding an exercise bout will be compared to the same meal on a baseline (no exercise) day and between the two exercise times.
Interstitial Glucose Concentration Variability | 3 days (1 day before to 1 day after exercise)
  Glucose will be charted using continuous glucose monitors. The day immediately before exercise will be used as baseline, the day of exercise to assess the acute response, and the day after exercise to assess lasting effects on glucose concentration variability.
Time Spent in Interstitial Glucose Concentration Range | 3 days (1 day before to 1 day after exercise)
  Glucose will be charted using continuous glucose monitors. The day immediately before exercise will be used as baseline, the day of exercise to assess the acute response, and the day after exercise to assess lasting effects on glycemic variability. Daily time spent in low (<3.9mmol/L), high (>10mmol/L) and within target glycemic range (3.9-10mmol/L) will be calculated on each occasion.
Nocturnal Interestitial Glucose Concentration | 2 days (day of, and 1 day after exercise)
  Glucose will be charted using continuous glucose monitors. The day immediately before exercise will be used as baseline, the day of exercise to assess the acute response, and the day after exercise to assess lasting effects on glycemic variability. Nocturnal glycemia (00:00-06:00) for each day will be compared on each exercise occasion.
Metabolic Response to Exercise | 1 hour (5 minutes before, 5 minutes after and 60 minutes after exercise)
  Changes in blood, skeletal muscle and subcutaneous adipose tissue metabolite levels will be assessed by broad-spectrum, untargeted metabolomics. Samples will be collected immediately before (-5 minutes) and after (+5 minutes) each exercise bout. An additional blood sample will be collected one hour after exercise completion (+60 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Wallberg-Henriksson, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data underlying results reported in a publication will be shared after deidentification.
Time Frame: Data will be made available indefinetly after publication.
Access Criteria: Data will be available for any purpose.

REFERENCES:
- [Derived] Keller MJ, Brady AJ, Smith JAB, Savikj M, MacGregor K, Jollet M, Oberg SB, Nylen C, Bjornholm M, Rickenlund A, Carlsson M, Caidahl K, Krook A, Pillon NJ, Zierath JR, Wallberg-Henriksson H. Inflammatory markers and blood glucose are higher after morning vs afternoon exercise in type 2 diabetes. Diabetologia. 2025 Sep;68(9):2023-2035. doi: 10.1007/s00125-025-06477-5. Epub 2025 Jun 28. PMID 40580209